CLINICAL TRIAL: NCT00584389
Title: The Effect of Rimonabant on Energy Expenditure, Fat Metabolism and Body Composition
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Suspension of licence for rimonabant by European Medicines Agency
Sponsor: University of Surrey (Other)
Collaborators: European Foundation for the Study of Diabetes (Other); Royal Surrey County Hospital NHS Foundation Trust (Other)
Responsible Party: Professor Margot Umpleby, University of Surrey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EC/2006/117/PGMS; Eudract 2006-006424-18
Record Dates: First submitted 2007-12-11; First posted 2008-01-02 (Estimated); Last update posted 2010-04-19 (Estimated); Status verified 2010-04

CONDITIONS: Obesity
Keywords: Obesity; Energy expenditure; Fatty acid; Triglyceride
MeSH Terms: conditions — Obesity | interventions — Rimonabant; Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Rimonabant treatment (20mg/d) for 12 weeks
  Interventions: Drug: rimonabant
- 2 (Other): Dietary intervention
  Interventions: Behavioral: Dietary intervention

INTERVENTIONS:
Drug: rimonabant — 20mg/d (oral) once daily for 12 weeks
  Other Names: Acomplia
  Arms: 1
Behavioral: Dietary intervention — Dietary intervention to match weight loss in group 1. The energy prescription will be based on the estimate of the energy deficit estimated from the weight loss in group one. For example a weight loss of 5kg over 12 weeks equates to an approximate energy deficit of 30,000 kcal or a daily energy reduction of approximately 357 kcal. If this is achieved in group 1 the daily energy target for subjects in group 2 will be daily energy expenditure minus 357 kcal.For the subjects randomised to the dietary intervention group there will be a delay until group 1 subjects have completed the study.
  Arms: 2

SUMMARY:
This study will determine in obese subjects the direct effects of the weight loss drug rimonabant (ie independent of weight loss) on energy expenditure, fat metabolism and and body fat distribution. We hypothesise that rimonabant will increase energy expenditure. The fuel for the increased energy expenditure will come from fat. As a result of burning more fat there will be a decrease in fat in blood and an improvement in the body's response to insulin.

DETAILED DESCRIPTION:
In obese subjects (BMI 33-38kg/m2) completing 12 months of treatment with the CB1 antagonist rimonabant (SR141716) there was an average weight loss from baseline of approximately 8.5 kg. These studies also showed the weight loss was accompanied by a decrease in plasma triglyceride (TG), an increase in HDL cholesterol and an improvement in insulin sensitivity measured by HOMA-IR. When adjusted for weight loss 50% of the improvements in TG, HDL cholesterol, and insulin sensitivity was not attributable to weight loss. This suggests that rimonabant has direct effects on fat metabolism.

This study will investigate the direct effects of rimonabant (ie independent of weight loss) in a 2 group randomised study. One group will receive rimonabant for 12 weeks and the other group will have a dietary intervention to match the weight loss in the rimonabant group. Measurements of energy expenditure (using indirect calorimetry and Actiheart monitors),fatty acid and triglyceride metabolism (using stable isotope techniques) and body fat distribution (by magnetic resonance imaging) will be made before and after the intervention. To determine the possible mechanisms of the changes in metabolism, gene expression of key regulators of fatty acid metabolism in adipose and muscle tissue and circulating levels of adipokines will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasian postmenopausal women
* BMI 30-38

Exclusion Criteria:

* Not currently weight-stable
* Diagnosed with diabetes
* Cardiovascular disease
* Endocrine disease
* Hepatic and renal disorders
* Neurological/psychological illness/history of depression
* Previous surgical procedures for weight loss
* Medications known to alter body weight or appetite
* β-blockers, fibrates and metformin
* Severe under-reporting of food intake based on a 4 day food diary

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-07; Primary Completion 2009-04 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
The direct effect of rimonabant on energy expenditure | 12 weeks

SECONDARY OUTCOMES:
Whole body fatty acid production and oxidation rate. | 12 weeks
Triglyceride synthesis and clearance rate. | 12 weeks
Whole body fat distribution. | 12 weeks
Adipose tissue and muscle mRNA levels of key regulators of fatty acid metabolism. | 12 weeks
Insulin sensitivity. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David L Russell-Jones, MBBS,MD,FRCP, Study Director — UK National Health Service; Margot Umpleby, BA, PhD, Principal Investigator — University of Surrey
Locations (1):
- Royal Surrey County Hospital, Guildford, Surrey, United Kingdom

REFERENCES:
- [Background] Despres JP, Golay A, Sjostrom L; Rimonabant in Obesity-Lipids Study Group. Effects of rimonabant on metabolic risk factors in overweight patients with dyslipidemia. N Engl J Med. 2005 Nov 17;353(20):2121-34. doi: 10.1056/NEJMoa044537. PMID 16291982
- [Background] Van Gaal LF, Rissanen AM, Scheen AJ, Ziegler O, Rossner S; RIO-Europe Study Group. Effects of the cannabinoid-1 receptor blocker rimonabant on weight reduction and cardiovascular risk factors in overweight patients: 1-year experience from the RIO-Europe study. Lancet. 2005 Apr 16-22;365(9468):1389-97. doi: 10.1016/S0140-6736(05)66374-X. PMID 15836887
- [Background] Pi-Sunyer FX, Aronne LJ, Heshmati HM, Devin J, Rosenstock J; RIO-North America Study Group. Effect of rimonabant, a cannabinoid-1 receptor blocker, on weight and cardiometabolic risk factors in overweight or obese patients: RIO-North America: a randomized controlled trial. JAMA. 2006 Feb 15;295(7):761-75. doi: 10.1001/jama.295.7.761. PMID 16478899
- [Derived] Backhouse K, Sarac I, Shojaee-Moradie F, Stolinski M, Robertson MD, Frost GS, Bell JD, Thomas EL, Wright J, Russell-Jones D, Umpleby AM. Fatty acid flux and oxidation are increased by rimonabant in obese women. Metabolism. 2012 Sep;61(9):1220-3. doi: 10.1016/j.metabol.2012.02.012. Epub 2012 Mar 24. PMID 22445512